CLINICAL TRIAL: NCT03153098
Title: Physical Activity Promotion in Areas of Deprivation for Inactive Adults With Cardiovascular Disease (CVD) Risk: An Evaluation of Active Herts
Brief Title: An Evaluation of the Active Herts Physical Activity Programme
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of East Anglia (Other)
Collaborators: University of Hertfordshire (Other); Hertfordshire Sports Partnership (Unknown); Sport England (Other); Broxbourne Borough Council (Unknown); East and North Hertfordshire Clinical Commisioning Group (Unknown); Hertfordshire Valley Clinical Commisioning Group (Unknown); Hertfordshire Public Health (Unknown)
Responsible Party: Sponsor
Other Study IDs: ActiveHerts
Record Dates: First submitted 2017-05-05; First posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Physical Activity
Keywords: physical activity; intervention; behaviour change; inactive adults; behaviour change techniques; well-being
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard delivery: Participants will receive a behaviour change technique booklet, consultations (baseline, and optional at 3, 6, and 12 months), a booster phone call (week 2), motivational text messages (weeks 3, 6, and 12), and signposting to 12 weeks of exercise classes.
  Interventions: Behavioral: Active Herts
- Enhanced delivery: Participants will receive the same as intervention but the 12 weeks of exercise will be free and tailored to their needs, and there will be optional exercise 'buddies' available.
  Interventions: Behavioral: Active Herts

INTERVENTIONS:
Behavioral: Active Herts — Active Herts is a community physical activity intervention aimed at inactive adults aged 16 and over who have one or more risk factors for CVD and/or a mild to moderate mental health condition. The programme uses the latest evidence-based behaviour change techniques to target physical activity, wellbeing, and key drivers of behaviour from the COM-B model of behaviour change.
  Other Names: Healthy and Active In Herts

SUMMARY:
There is a high prevalence of inactive adults in the United Kingdom (UK), many of whom suffer from conditions such as diabetes, cardiovascular disease, and poor mental health. These problems often co-exist more frequently in areas of higher socio-economic deprivation. There is an ongoing need to test the effectiveness, acceptability, and sustainability of community physical activity interventions. The Active Herts programme is a community physical activity programme aimed at inactive adults aged 16 and over who have one or more risk factors for cardiovascular disease (CVD) and/or a mild to moderate mental health condition. The programme uses the latest evidence-based behaviour change techniques to target physical activity, wellbeing, and key drivers of behaviour from the COM-B ('Capability', 'Opportunity', 'Motivation' and 'Behaviour') model of behaviour change.

This evaluation will follow a mixed-methods longitudinal (baseline, and 3, 6 and 12 month follow-ups) pragmatic observational design. Two types of programme are being delivered, each in a different area. In one, group participants will receive a behaviour change technique booklet, consultations (baseline, and optional at 3, 6, and 12 months), a booster phone call (week 2), motivational text messages (weeks 3, 6, and 12), and signposting to 12 weeks of exercise classes. In the other 'enhanced delivery' group, participants will receive the same but the 12 weeks of exercise will be free and tailored to their needs, and there will be optional exercise 'buddies' available. An outcome evaluation will assess changes in physical activity as the primary outcome, and sporting participation, sitting, wellbeing, psychological capability, and reflective motivation as secondary outcomes. A process evaluation will use both one-to-one interviews and focus groups to explore the views of stakeholders, delivery staff, and participants over three phases (set-up, deviations in the delivery of the intervention, and looking back over the intervention). Economic evaluation will examine the costs of the Active Herts programme against the benefits gained in terms of reduced risk of morbidity from a range of chronic conditions.

This study will measure key drivers of physical activity using up to date behaviour change theory, allowing evaluation of not only whether physical activity has increased but also why. The research will inform the future development of a scalable intervention that can be more robustly tested in a randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* inactive adults and do less than 30mins of physical activity per week
* aged 16 or over
* resident of Hertfordshire boroughs, including Broxbourne, Hertsmere, Stevenage or Watford

Referred patients and clients may also have:

* a long term medical condition such as type 2 diabetes, hypertension, high cholesterol etc.
* a mild to moderate mental health condition such as anxiety, depression or stress
* a history or family history of heart disease

Exclusion Criteria:

* participants not able to give informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will live in one of four Hertfordshire districts (Broxbourne, Stevenage, Hertsmere, and Watford), United Kingdom. The four districts contain the highest number of deprived Lower Super Output Areas (LSOA) in Hertfordshire and are in the five highest rates of under 75 mortality rate from CVD (2-3%), adult obesity (8-10%), and diabetes (4-6%). A life expectancy gap of 6-9.6 years exists between the most and least deprived areas across these districts. Less than 50% of this population participate in 30 minutes of physical activity once per week.
Sampling Method: Non-Probability Sample
Enrollment: 739 (Estimated)
Dates: Start 2016-01-07 (Actual); Primary Completion 2019-01-07 (Estimated); Study Completion 2019-01-07 (Estimated)

PRIMARY OUTCOMES:
Change in Physical activity from baseline | 12 months
  Assessed using the International Physical Activity Questionnaire (IPAQ)

SECONDARY OUTCOMES:
Change in mental well-being from baseline | Short term (3 months), longer term (6 and 12 months)
  Assessed using Warwick Edinburgh well-being scale
Change in perceptions of health from baseline | Short term (3 months), longer term (6 and 12 months)
  EuroQOL five dimensions questionnaire (EQ-5D)
Readiness to change behaviour | Short term (3 months), longer term (6 and 12 months)
  Key determinants of behaviour - measured using COM-B Capability, Opportunity, and Motivation

OTHER OUTCOMES:
Delivery fidelity | End February 2017, Summer 2017, Autumn 2018
  A process evaluation of Active Herts will take place in three phases with each phase exploring a different theme. Data will be collected in the form of one-to-one interviews with stakeholders, group interviews with the Get Active Specialists, and focus groups with participants. Stakeholders interviewed will include commissioners, higher intervention management, project delivery partners, and health service practitioners.
Programme cost-effectiveness | October 2017 - October 2018
  The economic evaluation will examine the costs of delivery of the Active Herts intervention against the benefits gained in terms of reduced risk of morbidity from a range of chronic conditions, the risk of which is associated with physical inactivity.

CONTACTS AND LOCATIONS:
Overall Officials: Andy Jones, Prof, Principal Investigator — University of East Anglia
Locations (1):
- University of East Anglia, Norwich, United Kingdom

REFERENCES:
- [Derived] Chater AM, Schulz J, Jones A, Burke A, Carr S, Kukucska D, Troop N, Trivedi D, Howlett N. Outcome evaluation of Active Herts: A community-based physical activity programme for inactive adults at risk of cardiovascular disease and/or low mental wellbeing. Front Public Health. 2022 Sep 9;10:903109. doi: 10.3389/fpubh.2022.903109. eCollection 2022. PMID 36159253
- [Derived] Howlett N, Jones A, Bain L, Chater A. How effective is community physical activity promotion in areas of deprivation for inactive adults with cardiovascular disease risk and/or mental health concerns? Study protocol for a pragmatic observational evaluation of the 'Active Herts' physical activity programme. BMJ Open. 2017 Nov 25;7(11):e017783. doi: 10.1136/bmjopen-2017-017783. PMID 29175885
- See also: Website for community intervention — http://www.activeherts.org.uk/